CLINICAL TRIAL: NCT01008462
Title: Sequential Autologous HCT / Nonmyeloablative Allogeneic HCT Using Related, HLA-Haploidentical Donors for Patients With High-Risk Lymphoma, Multiple Myeloma, or Chronic Lymphocytic Leukemia
Brief Title: Autologous Peripheral Blood Stem Cell Transplant Followed by Donor Bone Marrow Transplant in Treating Patients With High-Risk Hodgkin Lymphoma, Non-Hodgkin Lymphoma, Multiple Myeloma, or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2241.00; NCI-2009-01334 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2241.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: B-Cell Prolymphocytic Leukemia; Hypodiploidy; Loss of Chromosome 17p; Plasma Cell Leukemia; Progression of Multiple Myeloma or Plasma Cell Leukemia; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Childhood Hodgkin Lymphoma; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Plasma Cell Myeloma; Recurrent Small Lymphocytic Lymphoma; Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Non-Hodgkin Lymphoma; Refractory Plasma Cell Myeloma; Refractory Small Lymphocytic Lymphoma; t(14;16); t(4;14); T-Cell Prolymphocytic Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Prolymphocytic, B-Cell; Chromosome 17 deletion; Leukemia, Plasma Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia, Prolymphocytic, T-Cell; Waldenstrom Macroglobulinemia | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cyclophosphamide; Cytarabine; Etoposide; fludarabine phosphate; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (autologous HCT, donor HCT) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Autologous-Allogeneic Tandem Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Etoposide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo donor HCT
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo donor HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSC transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Procedure: Autologous-Allogeneic Tandem Hematopoietic Stem Cell Transplantation — Undergo autologous-donor tandem HCT
  Other Names: auto-allo HCT
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative study
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo donor HCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase II trial studies autologous peripheral blood stem cell transplant followed by donor bone marrow transplant in treating patients with high-risk Hodgkin lymphoma, non-Hodgkin lymphoma, multiple myeloma, or chronic lymphocytic leukemia. Autologous stem cell transplantation uses the patient's stem cells and does not cause graft versus host disease (GVHD) and has a very low risk of death, while minimizing the number of cancer cells. Peripheral blood stem cell (PBSC) transplant uses stem cells from the patient or a donor and may be able to replace immune cells that were destroyed by chemotherapy. These donated stem cells may help destroy cancer cells. Bone marrow transplant known as a nonmyeloablative transplant uses stem cells from a haploidentical family donor. Autologous peripheral blood stem cell transplant followed by donor bone marrow transplant may work better in treating patients with high-risk Hodgkin lymphoma, non-Hodgkin lymphoma, multiple myeloma, or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Event-free survival (EFS) at 1-year after autograft.

SECONDARY OBJECTIVES:

I. Relapse rates at 1-year after autograft.

II. Overall survival (OS) at 1-year after autograft.

III. Incidence of grades II-IV acute GVHD and chronic extensive GVHD.

IV. Non-relapse mortality (NRM) at 200 days and 1 year after allograft.

V. Donor engraftment at day +84.

VI. Incidence of infections.

OUTLINE:

CONDITIONING REGIMEN 1 (lymphoma, Waldenstrom macroglobulinemia, or chronic lymphocytic leukemia [CLL] with no dose limiting radiation or significant comorbidities: Patients receive cyclophosphamide intravenously (IV) on days -6 and -5. Patients undergo high-dose total body irradiation (TBI) twice daily (BID) on days -3 to -1.

CONDITIONING REGIMEN 2 (lymphoma, Waldenstrom Macroglobulinemia, CLL, with prior dose-limiting radiation, or significant comorbidities): Patients receive carmustine IV on day -7, etoposide IV BID on days -6 to -3, cytarabine IV BID on days -6 to -3, and melphalan IV on day -2.

CONDITIONING REGIMEN 3 (multiple myeloma or plasma cell leukemia, with no significant renal insufficiency or other significant comorbidities): Patients receive high-dose melphalan IV on day -2.

CONDITIONING REGIMEN 4 (multiple myeloma or plasma cell leukemia, with significant renal insufficiency or other significant comorbidities): Patients receive lessened dose of melphalan IV on day -2.

PBSC TRANSPLANTATION: All patients undergo autologous PBSC transplantation on day 0.

WAITING INTERVAL: Between 40 and 120 days.

NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV once daily (QD) on days -6 to -2 and cyclophosphamide IV QD on days -6 to -5 and day 3. Patients infused with donor's peripheral blood stem cells will additionally receive cyclophosphamide IV on day 4. Patients undergo low-dose TBI on day -1.

ALLOGENEIC BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.

GRAFT VERSUS HOST DISEASE PROPHYLAXIS: Beginning on day 4, patients receive tacrolimus orally (PO) or IV and taper beginning on day 86 if no graft-versus-host disease. Patients also receive mycophenolate mofetil PO thrice daily (TID) on days 4 - 35.

PERIPHERAL BLOOD COUNT SUPPORT: Patients receive filgrastim (G-CSF) IV or subcutaneously (SC) beginning from day 4 and continue till blood counts recover.

ALLOGENEIC PERIPHERAL BLOOD MONONUCLEAR CELLS (PBMC) TRANSPLANTATION: Patients undergo donor PBMC transplantation on day 0.

GRAFT VERSUS HOST DISEASE PROPHYLAXIS: Beginning on day 5, patients receive tacrolimus orally (PO) or IV and taper beginning on day 86 if no graft-versus-host disease. Patients also receive mycophenolate mofetil PO thrice daily (TID) on days 5 - 35.

PERIPHERAL BLOOD COUNT SUPPORT: Patients receive filgrastim IV or SC beginning from day 5 and continue till blood counts recover.

After completion of study treatment, patients are followed up annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have the capacity to give informed consent
* Detectable tumor prior to mobilization regimen
* Patients with stored autologous stem cells will be allowed
* Stem cells from an identical donor could be used for autologous hematopoietic cell transplant (HCT)
* Marrow is the preferred source of stem cells from the HLA-haploidentical donor, however, peripheral blood mononuclear cells (PBMC) could be used as stem cell source, after clearance with the Fred Hutchinson Cancer Research Center (FHCRC) principal investigator, in the case of difficulties or contraindications to bone marrow harvest from the donor
* Cross-over to other tandem autologous-allogeneic research protocol (#1409 or other appropriate protocol) will be allowed if a suitable HLA-matched related or unrelated donor is identified before receiving the allogeneic transplantation and if the patient meets the eligibility criteria of the subsequent study
* Cross-over from other tandem autologous-allogeneic research protocol (#1409 or other appropriate protocol) will be allowed if the patient loses the suitable HLA-matched related or unrelated donor but has an available HLA-haploidentical donor before receiving the allogeneic transplantation and if the patient meets the eligibility criteria of the subsequent study
* Lymphoma: patients with

  * Diagnosis of non-Hodgkin lymphoma (NHL) or Hodgkin's lymphoma (HL), of any histological grade
  * Refractory or relapsed disease after standard chemotherapy
  * High risk of early relapse following autograft alone
* Waldenstrom's macroglobulinemia: must have failed 2 courses of therapy
* CLL:

  * Patients with either a:

    * Diagnosis of T-cell CLL or T-cell prolymphocytic leukemia (PLL) who have failed initial chemotherapy, patients with T cell CLL or PLL or
    * Diagnosis of B-cell CLL, B-cell small lymphocytic lymphoma, or B-cell CLL that progressed to PLL who either:

      1. Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. 2-chlorodeoxyadenosine [CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine (or another nucleoside analog)
      2. Failed any aggressive chemotherapy regimen, such as fludarabine, cyclophosphamide and rituximab (FCR), at any time point
      3. Have "17p deletion" cytogenetic abnormality and relapsed at any time point after initial chemotherapy
  * Harvesting criteria for autologous HCT:

    * Previously collected PBMC may be used
    * Circulating CLL cells < 5000
  * Marrow involvement with CLL cells < 50%
* Multiple myeloma (MM): patients who

  * Have received induction therapy for a minimum of 4 cycles
  * In addition, patients must meet at least one of the following criteria I-IX (I-VII at time of diagnosis or pre-autograft):

    * Any abnormal karyotype by metaphase analysis except for isolated t(11,14),
    * Fluorescent in situ hybridization (FISH) translocation 4:14,
    * FISH translocation 14:16,
    * FISH deletion 17p,
    * Beta2 (B2)-microglobulin > 5.5 mg/ml,
    * Cytogenetic hypodiploidy
    * Plasmablastic morphology (>= 2%)
    * Recurrent or non-responsive (less than partial remission [PR]) MM after at least two different lines of conventional chemotherapy
    * Progressive MM after a previous autograft (provided stored autologous cluster of differentiation [CD]34 cells are available)
* Plasma cell leukemia: after induction chemotherapy
* DONOR: Related donors who are genotypically identical for one HLA haplotype and who may be mismatched at the HLA-A, -B, -C or DRB1 loci of the unshared haplotype with the exception of single HLA-A, -B or -C allele mismatches
* DONOR: Marrow is the preferred source of stem cells from the HLA-haploidentical donor, however PBMC could be used as stem cell source, after clearance with the FHCRC principal investigator, in the case of difficulties or contraindications to bone marrow harvest from the donor
* DONOR: In the case that PBMC will be used as stem cell source, ability of donors < 18 years of age to undergo apheresis without use of a vascular access device; vein check must be performed and verified by an apheresis nurse prior to arrival at the Seattle Cancer Care Alliance (SCCA)
* DONOR: Age >= 12 years of age

Exclusion Criteria:

* Life expectancy severely limited by disease other than malignancy
* Seropositive for the human immunodeficiency virus
* Female patients who are pregnant or breastfeeding
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years

  * This exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with fungal infection and radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Symptomatic coronary artery disease or ejection fraction < 40% or other cardiac failure requiring therapy (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Corrected diffusion capacity of the lungs for carbon monoxide (DLCO) < 50% of predicted, forced expiratory volume in one second (FEV1) < 50% of predicted, and/or receiving supplementary continuous oxygen; the FHCRC principal investigator (PI) of the study must approve of enrollment of all patients with pulmonary nodules
* Patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; the patient will be excluded if he/she is found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Karnofsky score < 50% for adult patients
* Lansky play-performance score < 40 for pediatric patients
* Patient with poorly controlled hypertension despite multiple antihypertensives
* DONOR: Donor-recipient pairs in which the HLA-mismatch is only in the host-versus-graft (HVG) direction
* DONOR: Infection with human immunodeficiency virus (HIV)
* DONOR: Weight < 20 kg
* DONOR: A positive anti-donor cytotoxic crossmatch

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sorror, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [15 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: Number of patients surviving without relapsed/progressive disease
Time Frame: 1 Year post-autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 16
Participants | 9

2. Secondary Outcome: Number of Patients With Relapsed/Progressive Disease
Description: Relapse/Progression defined as:
  Nodes, liver, and/or spleen ≥50% increased or new by physical exam / imaging studies.
  Circulating lymphocytes ≥50% increased by morphology and/or flow cytometry. Richter's transformation by lymph node biopsy .
Time Frame: 1 year post-autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 16
Participants | 6

3. Secondary Outcome: Overall Survival
Description: Number of patients surviving one year post-autograft
Time Frame: 1 year post-autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 16
Participants | 10

4. Secondary Outcome: Number of Patients With Grade II-IV Acute Graft-versus-Host-Disease and/or Chronic Extensive Graft-versus-Host-Disease
Description: aGVHD The diagnosis of aGVHD is identified through various stages and grading of the disease related to Skin (Rash), Gut (Diarrhea, Nausea/vomiting and/or anorexia) and the liver (Bilirubin) assessed by severity and grading scale outlined in the section Grafts vs Hosts by Sullivan (1999).
  GVHD Grades Grade I: 1-2 Skin Rash; No gut or liver involvement Grade II: Stage 1-3 Skin rash; Stage 1 gut and/or stage 1 liver involvement Grade III: Stage 2-4 gut involvement and/or stage 2-4 liver involvement with or without rash Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
  CGVHD The diagnosis of cGVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: 1 year post-allograft,
Population: Two patients are not evaluable for Graft-versus-Host-Disease due to disease progression; they failed the study and did not receive the allogeneic transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 14
Participants
  Acute Graft-versus-Host-Disease | 8
  Chronic extensive Graft-versus-Host-Disease | 1

5. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Number of patients with non-relapse mortalities.
Time Frame: 200 days and 1 Year post-allograft
Population: Two patients are not evaluable for GVHD due to disease progression; they failed the study and did not receive the allogeneic transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 14
Participants
  200 days | 0
  1 Year | 1

6. Secondary Outcome: Number of Patients Who Engrafted
Description: Number of patients with donor engraftment.
Time Frame: Day 84 post-allograft
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 14
Participants | 13

7. Secondary Outcome: Number of Patients Who Had Infections
Description: Number of patients who had infections.
Time Frame: 1 Year post-autograft
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Autologous HCT, Donor HCT)
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200; All-Cause Mortality: Conditioning through 1 Year.
Arm/Group | Treatment (Autologous HCT, Donor HCT)
All-Cause Mortality (participants affected / at risk) | 6/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Autologous HCT, Donor HCT) (N=16)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Autologous HCT, Donor HCT) (N=16)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3)
Fever (General disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT01008462/Prot_SAP_000.pdf